# Investigating Public Enthusiasm for Mammography Screening in Denmark

## Statistical Analysis Plan

NCT04509063 Unique Protocol ID: 2016-051-000001, 1835

Date: January 11, 2021

## Statistical Analysis Plan

#### Description of data

 Table with prevalence of women with an irrational preference for hypothetical screening test (willing to participate in screening with no benefits only harms). In addition, prevalences will be estimated for sub-groups based on what women said they read and believed about the screening test reducing breast cancer mortality or not (two different questions).

### Logistic regression

- Univariate logistic regression will be used to investigate different variables' impact
  on willingness to participate in hypothetical screening test. This will be conducted as
  a univariate correction due to low sample size (lower participation rate than
  anticipated).
- The analysis will be corrected for each of the following variables: age, health literacy level, education, civil status, economy, municipality, information on whether a participant is immigrant, descendent or of Danish origin, previous breast cancer diagnosis, perceived risk of developing breast cancer, worry about breast cancer, close family/friends with breast cancer, and perceived riskiness of hypothetical screening test.
- In a sensitivity analysis, the impact of decision certainty will be investigated (How certain are you about your previous answer (that you would participate/would not participate? Answered on 7-point Likert scale)).

Note: The original plan for the main analysis was to compare the two groups of women randomized to different information groups (detailed vs. non-detailed information about the harms of screening). However, due to lower participation rate and therefore smaller sample size than expected, information group was disregarded in the main analysis. The two groups will still be compared in a secondary analysis (the investigator will be blinded for group assignment). This decision was made before getting access to data from the questionnaire.